CLINICAL TRIAL: NCT04308148
Title: Does Medical Cannabis Reduce Opioid Use in Adults With Pain: An Observational Study
Brief Title: Does Medical Cannabis Reduce Opioid Use in Adults With Pain
Acronym: ReLeaf-E
Status: Completed | Type: Observational
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: Laura and John Arnold Foundation (Other); Vireo Health (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-10029
Record Dates: First submitted 2020-03-12; First posted 2020-03-13 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Opioid Use; Marijuana; Chronic Pain
Keywords: Opioid; Marijuana; Cannabis; Pain
MeSH Terms: conditions — Marijuana Abuse; Chronic Pain; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study will examine how medical cannabis use affects opioid analgesic use. This landmark study will be among the first to examine the effect of medical cannabis with different THC/CBD (Tetrahydrocannibinol/Cannabidiol) content on opioid use as well as adverse events.

DETAILED DESCRIPTION:
This study will examine how medical cannabis use affects opioid analgesic use, with particular attention to THC/CBD (Tetrahydrocannibinol/Cannabidiol) content and adverse events. We will enroll adults with (a) severe or chronic neuropathic or joint pain, (b) prescribed opioid analgesic use, (c) active certification for medical cannabis, and (d) intends to have soft gel capsule products dispensed at Vireo (medical cannabis dispensary) (including a high THC:low CBD product, an equal THC:CBD (Tetrahydrocannibinol:Cannabidiol) product, and a low THC:high CBD product). Over the 14 weeks, data sources will include questionnaires; medical, pharmacy, and Prescription Monitoring Program (PMP) records; and urine samples. The primary independent variable will be type of soft gel capsule product, and the primary outcome will be cumulative opioid analgesic dose.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* English or Spanish fluency
* Actively certified for medical cannabis
* Intends to have a soft-gel capsule product dispensed at Vireo
* Medical cannabis qualifying conditions or complications of "chronic or severe pain" or "pain that degrades health and functional capability as an alternative to opioid use or substance use disorder"
* Joint or neuropathic pain
* Current severe pain
* Dispensed opioid analgesics within the last 60 days

To maintain the integrity of the study, we do not disclose all inclusion criteria to potential participants.

Exclusion Criteria:

* Inability to provide informed consent
* Inability to complete study visits over 14 weeks
* Terminal illness
* Current or prior psychotic disorder
* Buprenorphine or methadone treatment for opioid use disorder within the past year
* Allergies to tapioca or coconut
* Currently pregnant, planning to become pregnant within the next 3 months, or breastfeeding
* Condition that is considered by a pharmacist or medical provider to be a contraindication to medical cannabis use (e.g. unstable cardiac arrhythmia or specific drug-use interaction)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with chronic pain, who are taking opioids and are actively certified for medical cannabis in New York.
Sampling Method: Non-Probability Sample
Enrollment: 217 (Actual)
Dates: Start 2020-10-06 (Actual); Primary Completion 2024-03-13 (Actual); Study Completion 2024-03-13 (Actual)

PRIMARY OUTCOMES:
Opioid analgesic use | Opioid analgesic use will be weekly cumulative dose of opioid analgesics over 14 weeks.
  The primary outcome will be opioid analgesic use.

SECONDARY OUTCOMES:
Adverse events | Adverse events will be over 14 weeks
  (e.g. Cannabis use disorder, illicit drug use, diversion of medical cannabis, accidents and injuries)

CONTACTS AND LOCATIONS:
Overall Officials: Julia Arnsten, MD, MPH, Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- Montefiore Health System, The Bronx, New York, United States